CLINICAL TRIAL: NCT06376604
Title: Use of a Fasting Mimicking Diet in Patients Undergoing Chemotherapy for Gynecologic Malignancies
Brief Title: Fasting Mimicking Diet in Chemotherapy of Gynecologic Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: L-Nutra Inc (Industry)
Collaborators: University of Tennessee Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LNT55
Record Dates: First submitted 2024-04-11; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cancer, Ovarian; Chemotherapy Effect; Calorie Deficiency; Fasting, Intermittent
Keywords: Fasting mimicking diet; Gynecologic malignancy; Chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Intermittent Fasting | interventions — Drug Therapy

STUDY DESIGN:
Masking Description: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMD (Experimental): In addition to the standard care, subject will consume a 5-day fasting mimicking diet.
  Interventions: Other: Fasting Mimicking Diet; Drug: Chemotherapy
- Control (Active Comparator): Subjects will receive the standard care and no dietary changes.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Other: Fasting Mimicking Diet — Subject will consume 6 cycles of 5-day fasting mimicking diet: 3 days prior to, the day of, and 1 day following chemotherapy treatments.
  Arms: FMD
Drug: Chemotherapy — 6 cycles of standard chemotherapy for the gynecologic malignancy.

SUMMARY:
This study evaluates how lifestyle modifications that may be made to manage chemotherapy side effects in patients with gynecologic malignancies.

DETAILED DESCRIPTION:
Since chemotherapy remains one of the primary treatment modalities for gynecologic malignancies, there is increasing interest in non-pharmacological methods of reducing chemotherapy side effects in cancer patients. Our goal is to increase the knowledge surrounding lifestyle modifications, specifically the fasting mimicking diet, on chemotherapy-related side effects, which may be more acceptable to patients than a previously studied water-only fasting diet. To expand this knowledge, The investigators will focus on patients undergoing chemotherapy for gynecologic malignancies. These patients will be assigned to no dietary restriction (control group) or a 5-day fasting mimicking diet (FMD by L-Nutra) for three days prior to, the day of, and one day following chemotherapy treatments (treatment group). The investigators aim to evaluate the feasibility of a fasting mimicking diet in addition to its metabolic effects on the body, patient reported side effects, patient quality of life, deviations or delays in treatment plans, and hospital admissions. Our hypothesis is that a fasting mimicking diet will significantly decrease chemotherapy-related side effects while providing good quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 35-70 years old (both inclusive)
* Biopsy proven gynecologic malignancy
* Scheduled to or currently undergoing chemotherapy, with a minimum of 6 cycles remaining
* BMI greater than or equal to 18.5
* Adequate renal function (serum creatinine less than 1.5 times the upper limit of normal)
* Willing to adhere to a 5-day fasting mimicking diet

Exclusion Criteria:

* Pregnant or nursing mothers
* Prisoners
* Patients with diabetes or history of hypoglycemia
* Taking daily medications that cannot be safely taken without food
* History of significant or unstable cardiac disease such as congestive heart failure or history of myocardial infarction, stroke or pulmonary embolism within the last 3 months, renal failure, history of - eating disorder, dementia, psychosis, impaired physical mobility.
* Significant medical comorbidity that would be dangerous with a fasting mimicking diet.
* Any known or suspected food allergies that overlap with the FMD/Transitional diet by L-Nutra meal kit ingredients.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study focuses on the chemotherapy of gynecologic malignancies.
Enrollment: 30 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life by National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy Ovarian Cancer Symptom Index (NFOSI-18) questionnaire | Week 0-21
  The NFOSI-18 questionnaire allows for a uniform assessment of health-related quality of life through an 18-question (5-point Likert-type scale) survey including four subscale domains: Disease-Related Symptoms - Physical, Disease-Related Symptoms - Emotional, Treatment Side Effects. and Function/Well-Being. To calculate subscale scores, sum the item scores within each domain. Higher subscale scores indicate more significant symptom burden or impact. The total score is obtained by summing all 18 item scores. A higher total score reflects more severe symptoms overall.
Rate of Adherence | Week 0-21
  The ability to adhere to a 5-day fasting mimicking diet.

SECONDARY OUTCOMES:
Change in Body Weight | Week 0, Week12, Week 21
  Change in body weight.
Change in Body Composition | Week 0, Week12, Week 21
  Changes in weight, skeletal muscle mass, body fat percentage by the Inbody(R) Body Composition Analyzer.
Change in HbA1c | Week 0, Week 21
  Change in blood HbA1c.
Change in Insulin Like Growth Factor 1 (IGF-1) Concentration | Week 0, Week 21
  Change in blood insulin like growth factor 1 level.
Change in Fasting Insulin Concentration | Week 0, Week 21
  Change in fasting insulin level.
Change in Fasting Glucose Concentration | Week 0, Week 21
  Change in fasting glucose level.
Change in High-sensitivity C reactive protein Concentration | Week 0, Week 21
  Change in blood C reactive protein level.
Change in Leptin Concentration | Week 0, Week 21
  Change in blood leptin level.
Change in planned chemotherapy regimen | Week 0-21
  Deviation from the planned chemotherapy regimen.
Number of Hospitalization Days | Week 0-21
  Days of hospitalization
Rate of Chemotherapy Side Effects | Week 0-21
  Rate of Adverse effects associated with chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Boone, Principal Investigator — The University of Tennessee Medical Center
Locations (1):
- The University of Tennessee Medical Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caffa I, Spagnolo V, Vernieri C, Valdemarin F, Becherini P, Wei M, Brandhorst S, Zucal C, Driehuis E, Ferrando L, Piacente F, Tagliafico A, Cilli M, Mastracci L, Vellone VG, Piazza S, Cremonini AL, Gradaschi R, Mantero C, Passalacqua M, Ballestrero A, Zoppoli G, Cea M, Arrighi A, Odetti P, Monacelli F, Salvadori G, Cortellino S, Clevers H, De Braud F, Sukkar SG, Provenzani A, Longo VD, Nencioni A. Fasting-mimicking diet and hormone therapy induce breast cancer regression. Nature. 2020 Jul;583(7817):620-624. doi: 10.1038/s41586-020-2502-7. Epub 2020 Jul 15. PMID 32669709
- [Background] de Groot S, Lugtenberg RT, Cohen D, Welters MJP, Ehsan I, Vreeswijk MPG, Smit VTHBM, de Graaf H, Heijns JB, Portielje JEA, van de Wouw AJ, Imholz ALT, Kessels LW, Vrijaldenhoven S, Baars A, Kranenbarg EM, Carpentier MD, Putter H, van der Hoeven JJM, Nortier JWR, Longo VD, Pijl H, Kroep JR; Dutch Breast Cancer Research Group (BOOG). Fasting mimicking diet as an adjunct to neoadjuvant chemotherapy for breast cancer in the multicentre randomized phase 2 DIRECT trial. Nat Commun. 2020 Jun 23;11(1):3083. doi: 10.1038/s41467-020-16138-3. PMID 32576828
- [Background] Finnell JS, Saul BC, Goldhamer AC, Myers TR. Is fasting safe? A chart review of adverse events during medically supervised, water-only fasting. BMC Complement Altern Med. 2018 Feb 20;18(1):67. doi: 10.1186/s12906-018-2136-6. PMID 29458369
- [Background] Goncalves MD, Cantley LC. A 'fast'er way to treat breast cancer. Nat Metab. 2020 Jul;2(7):559-560. doi: 10.1038/s42255-020-0225-6. No abstract available. PMID 32694797
- [Background] Lee C, Raffaghello L, Brandhorst S, Safdie FM, Bianchi G, Martin-Montalvo A, Pistoia V, Wei M, Hwang S, Merlino A, Emionite L, de Cabo R, Longo VD. Fasting cycles retard growth of tumors and sensitize a range of cancer cell types to chemotherapy. Sci Transl Med. 2012 Mar 7;4(124):124ra27. doi: 10.1126/scitranslmed.3003293. Epub 2012 Feb 8. PMID 22323820
- [Background] Raffaghello L, Safdie F, Bianchi G, Dorff T, Fontana L, Longo VD. Fasting and differential chemotherapy protection in patients. Cell Cycle. 2010 Nov 15;9(22):4474-6. doi: 10.4161/cc.9.22.13954. Epub 2010 Nov 15. PMID 21088487
- [Background] Safdie FM, Dorff T, Quinn D, Fontana L, Wei M, Lee C, Cohen P, Longo VD. Fasting and cancer treatment in humans: A case series report. Aging (Albany NY). 2009 Dec 31;1(12):988-1007. doi: 10.18632/aging.100114. PMID 20157582
- [Background] Moss HA, Havrilesky LJ. The use of patient-reported outcome tools in Gynecologic Oncology research, clinical practice, and value-based care. Gynecol Oncol. 2018 Jan;148(1):12-18. doi: 10.1016/j.ygyno.2017.11.011. Epub 2017 Nov 23. PMID 29174565